CLINICAL TRIAL: NCT00265629
Title: A Clinical Investigation of Radiofrequency Ablation for the Treatment of Atrial Fibrillation Using the High Density Mesh Bard Ablation System
Brief Title: RF Ablation of Atrial Fibrillation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BEP-4405
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): RF ablation
  Interventions: Device: RF catheter ablation

INTERVENTIONS:
Device: RF catheter ablation — RF ablation using mesh device

SUMMARY:
This is an early feasibility trial designed to demonstrate whether a new ablation device can be used safely and effectively in treating atrial fibrillation.

This study is a prospective, nonrandomized, single-arm, multi-center trial to be conducted at a single study site

DETAILED DESCRIPTION:
This study is intended to evaluate the safety and preliminary effectiveness of the RFMesh BAS for electrophysiological mapping and radiofrequency ablation in the region of the ostium of a targeted pulmonary vein in the treatment of drug refractory paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are between 18 & 85 years of age.
2. Patients with a minimum of 2 episodes of symptomatic PAF within the last 6 months prior to baseline evaluation. At least one of these episodes must have been documented. Documentation may include electrocardiogram (ECG), trans telephonic monitoring (TTM), Holter monitoring (HM), or telemetry strip. Additional PAF episodes (i.e., verbal accounts from the patient) will be documented in the patient's study record.
3. Patients who have failed at least 1 class I or class III anti-arrhythmic medication regimen.
4. Patients with the ability to understand the requirements of the study, who have provided written informed consent and agreed to the study restrictions and to return for the required follow-up assessments.

Exclusion Criteria:

1. Any previous ablation of the left atrium (surgical or catheter based).
2. Permanent or persistent atrial fibrillation.
3. Recent myocardial infarction within 2 months
4. Currently unstable angina.
5. Any cardiac surgery during the previous 3 months.
6. Currently documented intracardiac thrombus by transesophageal echocardiography (TEE).
7. A left atrium > 50mm in major dimension.
8. A common ostium larger than 25 mm in major axis or any individual pulmonary vein larger than 25 mm in major axis.
9. Permanent leads in or through the right atrium.
10. Clinically significant valvular heart disease or a replacement heart valve.
11. Congestive heart failure (NYHA classification III or IV).
12. An ejection fraction <35%.
13. A contraindication to warfarin.
14. A contraindication to transseptal procedure.
15. Any cerebral ischemic event, including any transient ischemic attack (TIA), in the preceding 6 months.
16. Any known bleeding disorder.
17. Women who are known to be pregnant or nursing.
18. Uncontrolled hyperthyroidism.
19. Patients currently enrolled in any other clinical investigation.
20. Any other significant uncontrolled or unstable medical condition.
21. A life expectancy of less than one year.
22. Currently taking amiodarone or have taken amiodarone within 4 months prior to baseline evaluation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-08; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of the HDMA when used to map & ablate patients with AF, by assessing MCs at 7-days & 30 days post-procedure & assessing the occurrence of pulmonary vein stenosis at 3 & 12 months post-procedure. | 12 months
Evaluate the preliminary effectiveness of the HDMA when used to map and ablate patients with paroxysmal AF, by assessing APS & the freedom from recurrence of symptomatic AF at 3, 6 & 12 months post- procedure. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- David Haines, MD, Royal Oak, Michigan, United States